CLINICAL TRIAL: NCT02629172
Title: Drug Use Results Survey in Patients Infected With Hepatitis C Virus Genotype 1
Brief Title: Drug Use-results Survey in Patients Infected With Hepatitis C Virus Genotype 1
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-336
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Chronic Hepatitis C Virus
Keywords: Hepatitis C Virus (HCV); Paritaprevir; Ombitasvir; Ritonavir; Genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic infection of hepatitis C virus (HCV) Genotype 1 (GT1): Participants with confirmed chronic hepatitis C genotype 1, receiving paritaprevir/ritonavir/ombitasvir according to standard of care and in line with the current local label

SUMMARY:
The main objective of this study is to evaluate the safety and effectiveness of paritaprevir/ritonavir/ombitasvir used for patients infected with HCV genotype 1 in daily practice in Japan.

ELIGIBILITY:
Inclusion Criteria:

* HCV genotype 1 patients treated with paritaprevir/ritonavir/ombitasvir in daily practice

Exclusion Criteria:

* Patients who have been previously treated with paritaprevir/ritonavir/ombitasvir

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic Hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 3043 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Sustained Virologic Response (SVR12) | 12 weeks after the last dose of study drug
  Hepatitis C virus ribonucleic acid less than the lower limit of quantification 12 weeks after the last dose of study drug.

SECONDARY OUTCOMES:
Percentage of Participants with Virologic Failure After Treatment | Post-treatment 24 weeks
  Confirmed quantifiable hepatitis C virus ribonucleic acid (HCV RNA) at the end of 12 week treatment but subsequent viremia with HCV RNA greater than or equal to the lower limit of quantitation during follow-up period of 24 weeks after treatment.
Percentage of Participants with Sustained Virologic Response (SVR24) | 24 weeks after the last dose of study drug
  Hepatitis C virus ribonucleic acid less than the lower limit of quantification 24 weeks after the last dose of study drug.
Percentage of Participants with Virologic Failure During Treatment | Up to Week 12
  HCV RNA levels reach less than the lower limit of quantitation (LLOQ), then increase to greater than or equal to the LLOQ at any point during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (388):
- Japan (388):
  - Aichi Medical University Hosp /ID# 152220, Nagakute, Aichi-ken
  - Nagoya City University Hospital /ID# 153642, Nagoya, Aichi-ken
  - Japanese Red Cross Narita Hosp /ID# 155894, Narita-shi, Chiba
  - Kikkoman General Hospital /ID# 152139, Noda, Chiba
  - Matsuyama Red Cross Hosp /ID# 152271, Matsuyama, Ehime
  - NHO Kyushu Medical Center /ID# 153001, Fukuoka, Fukuoka
  - Fukuoka University Hospital /ID# 152272, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 152099, Kurume-shi, Fukuoka
  - Gifu University Hospital /ID# 152993, Gifu, Gifu
  - Kusunoki Hospital /ID# 152072, Fujioka, Gunma
  - Gunma University Hospital /ID# 154669, Maebashi, Gunma
  - National Hospital Organization Takasaki General Medical Center /ID# 152971, Takasaki-shi, Gunma
  - Fukuyama City Hospital /ID# 152322, Fukuyama-shi, Hiroshima
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 152165, Sapporo, Hokkaido
  - Sapporo Medical Univ Hosp /ID# 152992, Sapporo, Hokkaido
  - Kobe University Hospital /ID# 153004, Kobe, Hyōgo
  - The Hospital of Hyogo College of Medicine /ID# 157482, Nishinomiya-shi, Hyōgo
  - JA Toride Medical Center /ID# 153657, Toride, Ibaraki
  - Kanazawa University Ho /ID# 152174, Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital /ID# 152076, Morioka, Iwate
  - Nanpuh Hospital /ID# 153008, Kagoshima, Kagoshima-ken
  - Shonan Fujisawa Tokushukai Hospital /ID# 152967, Fujisawa-shi, Kanagawa
  - Shonan Kamakura General Hospital /ID# 152070, Kamakura-shi, Kanagawa
  - Yokohama City Univ Medical Ctr /ID# 153643, Yokohama, Kanagawa
  - Yokohama City University Hospital /ID# 154663, Yokohama, Kanagawa
  - Yokohama Municipal Citizen's Hospital /ID# 152151, Yokohama, Kanagawa
  - Kumamoto Shinto General Hospital /ID# 152149, Kumamoto, Kumamoto
  - Kyoto Prefect Univ Med /ID# 152236, Kyoto, Kyoto
  - Kyoto Prefect Univ Med /ID# 152981, Kyoto, Kyoto
  - JP Red Cross Kyoto Daiichi Hos /ID# 152221, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 152980, Sendai, Miyagi
  - Shinshu University Hospital /ID# 153632, Matsumoto-shi, Nagano
  - Nagasaki University Hospital /ID# 152233, Nagasaki, Nagasaki
  - Okayama University Hospital /ID# 152287, Okayama, Okayama-ken
  - Kansai Medical University Hospital /ID# 152269, Hirakata-shi, Osaka
  - Osaka Saiseikai Nakatsu Hospital /ID# 155967, Osaka, Osaka
  - Osaka Red Cross Hospital /ID# 152190, Osaka, Osaka
  - Osaka City University Hospital /ID# 152160, Osaka, Osaka
  - Nippon Life Saiseikai Public Interest Foundation Nippon Life Hospital /ID# 152279, Osaka, Osaka
  - Osaka Medical College Hospital /ID# 152307, Takatsuki -shi, Osaka
  - Saitama Medical Center, Saitama Medical University /ID# 153641, Kawagoe-shi, Saitama
  - Shiga Univ Med Science Hosp /ID# 153628, Ōtsu, Shiga
  - Hamamatsu University Hospital /ID# 154651, Hamamatsu, Shizuoka
  - Shizuoka General Hospital /ID# 152162, Shizuoka, Shizuoka
  - Jichi Medical University Hospital /ID# 152069, Shimotsuke-shi, Tochigi
  - Tokushima University Hospital /ID# 159455, Tokushima, Tokushima
  - Tokyo Teishin Hospital /ID# 157457, Chiyoda-ku, Tokyo
  - Tokyo Jikei Daisan Hospital /ID# 155896, Komae-shi, Tokyo
  - Kyorin University Hospital /ID# 152990, Mitaka-shi, Tokyo
  - Japanese Red Cross Medical Center /ID# 152219, Shibuya-ku, Tokyo
  - Showa University Hospital /ID# 153618, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 152288, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 152290, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 156383, Shinjuku-ku, Tokyo
  - Yamagata University Hospital /ID# 154664, Yamagata, Yamagata
  - University of Yamanashi Hospital /ID# 152164, Chuo-shi, Yamanashi
  - Ageo Central General Hospital /ID# 153002, Ageo
  - Sangane Clinic /ID# 162885, Aichi
  - Banbuntane Hotokukai Hospital /ID# 160909, Aichi
  - Masuda Family Clinic /ID# 155961, Aki-takata
  - Akita Kousei Medical Center /ID# 152183, Akita
  - Takahashi Naika /ID# 162888, Amagasaki
  - Kansai Rosai Hospital /ID# 152239, Amagasaki
  - Ikeda Hospital /ID# 152135, Amagasaki
  - Kato Michio Hepatology Clinic /ID# 152138, Amagasaki, Hyogo
  - Aomori Prefectural Central Hos /ID# 161749, Aomori
  - Konoe Hospital /ID# 158066, Arao
  - Japanese Red Cross Asahikawa /ID# 153552, Asahikawa
  - Asakura Medical Association Ho /ID# 152999, Asakura
  - Azumino Red Cross Hospital /ID# 160801, Azumino
  - Chiba Aoba Municipal Hospital /ID# 153016, Chiba
  - Chiba University Hospital /ID# 152988, Chiba
  - NHO Chiba-East-Hospital /ID# 152217, Chiba
  - Saisei Hospital /ID# 152277, Chiba
  - Fujishima Clinic /ID# 152216, Chiba
  - Seirei Sakura Citizen Hospital /ID# 152296, Chiba
  - Aioi Clinic /ID# 150059, Chichibu
  - Shonan Ishiguro Clinic /ID# 165272, Chigasaki
  - Shonan Tobu Sogo Hospital /ID# 152979, Chigasaki
  - Chikugo City Hospital /ID# 152318, Chikugo
  - Chitose City Hospital /ID# 156386, Chitose-shi
  - MIne Internal Medicine Clinic /ID# 155885, Fuchū
  - Tama Medical Center /ID# 158101, Fuchū
  - Fuji City General Hospital /ID# 159456, Fuji
  - Fukuchiyama City Hospital /ID# 157455, Fukuchiyama
  - Fukui Prefectural Hospital /ID# 152137, Fukui
  - Fukui Prefectural Hospital /ID# 152976, Fukui
  - University of Fukui Hospital /ID# 152169, Fukui
  - Tanaka Internal Medical Clinic /ID# 157499, Fukui
  - Hopsital of the University of Occupational and Enviromental Health /ID# 152998, Fukuoka
  - Saiseikai Fukuoka General Hosp /ID# 152167, Fukuoka
  - Fukuoka City Med Assoc Hosp /ID# 164143, Fukuoka
  - Shimizu Clinic /ID# 152166, Fukuoka
  - Chihaya Hospital /ID# 152223, Fukuoka
  - Fukushima Med Univ Hosp /ID# 154735, Fukushima
  - Clinic21 /ID# 153554, Fukushima
  - Rai Clinic /ID# 164133, Fukushima
  - Ishikawa Clinic /ID# 161747, Fukuyama
  - Morichika Internal Medicine /ID# 162887, Fukuyama
  - Gifu Municipal Hospital /ID# 152283, Gifu
  - Haramachi Red Cross Hospital /ID# 157447, Gunma
  - Hospital Hakodate Hokkaido /ID# 159457, Hakodate
  - Matsuda Internal Medicine /ID# 165064, Hamamatsu-shizuoka
  - Handa City Hospital /ID# 152140, Handa-shi
  - Mashiba Clinic /ID# 152097, Hannō
  - Hashima City Hospital /ID# 154658, Hashima
  - JA Hiroshima General Hospital /ID# 154729, Hatsukaichi
  - Higashihiroshima Medical Ctr /ID# 152970, Higashihiroshima
  - Mito Medical Center /ID# 154652, Higashiibaraki-gun
  - Higashiomicity Notogawa Hosp /ID# 152075, Higashiomi, Shiga
  - Wakakusa Daiichi Hospital /ID# 152201, Higashiosaka
  - Higashiosaka City General Hosp /ID# 153630, Higashiosaka-shi
  - Higashi-Omi Keiai Hospital /ID# 164954, Higashiōmi
  - Kousei Hospital /ID# 152159, Himeji
  - Kajihara Clinic /ID# 159451, Hiratsuka
  - Nakahata Gastroenterology Clin /ID# 164134, Hirosaki
  - Hirosaki University Hospital /ID# 153633, Hirosaki-aomori
  - Hiroshima Red Cross Hosp Atomi /ID# 152098, Hiroshima
  - Nishihara Nakamura Med Clinic /ID# 155999, Hiroshima
  - Hiroshima University Hospital /ID# 152319, Hiroshima
  - Hiroshima-Nishi Medical Center /ID# 161744, Hiroshima
  - Hiroshima Clinic /ID# 153614, Hiroshima
  - Hiroshima General Hosp W JP /ID# 152077, Hiroshima
  - Iwao Hospital /ID# 152306, Hita
  - Hitachi, Ltd., Hitachi Gen Hos /ID# 161748, Hitachi
  - Naganuma Municipal Hospital /ID# 152991, Hokkaido
  - Japanese Red Cross Kitami Hosp /ID# 153010, Hokkaido
  - Akashi City Hospital /ID# 150058, Hyōgo
  - Ashiya Municipal Hospital /ID# 150054, Hyōgo
  - Hyogo Prefectural Awaji Hosp /ID# 152237, Hyōgo
  - Hyogo Prefectural Kakogawa Med /ID# 152280, Hyōgo
  - Tokyo Dental College Ichikawa /ID# 154665, Ichikawa-shi
  - Iizuka Hospital /ID# 152186, Iizuka
  - Ikeda Municipal Hospital /ID# 152170, Ikeda
  - Nagasaki Prefecture Iki Hospit /ID# 154674, Iki
  - Nara Hosp Kinki Uni Fac Of Med /ID# 155895, Ikoma
  - Saiseikai Imabari Hospital /ID# 158100, Imabari
  - Ina Central Hospital /ID# 152144, Ina
  - Tokyo Med Uni Ibaraki Med Ctr /ID# 152121, Inashiki
  - Inuyama Chuo General /ID# 154672, Inuyama
  - Saitama Medical University Hos /ID# 152073, Iruma-gun
  - Saitama Medical University Hos /ID# 153616, Iruma-gun
  - Ise Red Cross Hospital /ID# 154670, Ise
  - Yamada Internal Medicine Clini /ID# 154786, Isesaki
  - Katakai Clinic /ID# 152163, Isesaki
  - Yawata Medical Center /ID# 152215, Ishikawa
  - Matto Ishikawa Public Hospital /ID# 153638, Ishikawa
  - Kamiiwade Internal Med-Neuro /ID# 160802, Iwade
  - Iwaki Kyoritsu General Hosp /ID# 153617, Iwaki
  - Yoshioka Clinic /ID# 152305, Iwaki
  - Nishimi Medical Clinic /ID# 161752, Iwakuni
  - Kayanoki Internal Medicine Cli /ID# 152235, Izumiōtsu
  - Juntendo Univ Shizuoka Hosp /ID# 153615, Izunokuni-shi
  - Kawabata Internal Medicine Gas /ID# 153629, Joetsu-niigata
  - Mitoyo General Hospital /ID# 152185, Kagawa
  - Konan Kakogawa Hospital /ID# 158102, Kakogawa
  - Yoshii Internal Medicine /ID# 158067, Kaminoyama
  - Kiyokawa Hospital /ID# 152156, Kanagawa
  - Nagase Medical Clinic /ID# 157498, Kanagawa
  - Hiratsuka City Hospital /ID# 154730, Kanagawa
  - Niwa Hospital /ID# 154762, Kanagawa
  - Fuji Clinic /ID# 152968, Kan’onjichō
  - Fujise Internal Medicine Clini /ID# 155886, Kashiwa
  - The Jikei Univ. Kashiwa Hosp. /ID# 152281, Kashiwa-shi
  - Fukuoka Tokushukai Medical Ctr /ID# 154654, Kasuga-shi
  - Kawase Clinic /ID# 152969, Kasugai
  - Sakamoto Internal Med Clinic /ID# 161745, Katori
  - Sekishindo Hospital /ID# 154653, Kawagoe
  - Saiseikai Kawaguchi Gen. Hosp. /ID# 153631, Kawaguchi-saitama
  - Kawasaki Municipal Tama Hospit /ID# 152132, Kawasaki
  - St. Marianna Univ Hospital /ID# 152218, Kawasaki
  - Kanto Rosai Hospital /ID# 152202, Kawasaki-shi, Kanagawa
  - Nakano Clinic /ID# 165262, Kazuno
  - Kirishima Medical Center /ID# 152095, Kirishima
  - Kojima Clinic /ID# 152285, Kiryū
  - Kimitsu Chuo Hospital /ID# 152995, Kisarazu
  - Kawazoe Internal Medicine Clin /ID# 154789, Kishima-gun
  - Kishiwada Tokushukai Hospital /ID# 165260, Kishiwada, Osaka
  - JR Kyushu Hospital /ID# 152074, Kitakyushu
  - Kokura Kinen Hospital /ID# 152997, Kitakyushu
  - Iwamoto Internal Medical Clini /ID# 152994, Kitakyushu
  - Kitasato University Medical Ce /ID# 150053, Kitamoto
  - Kobe City Medical Center West /ID# 152304, Kobe
  - Kobe City Medical Center West /ID# 153005, Kobe
  - Kobe Asahi Hospital /ID# 152173, Kobe
  - Kochi Red Cross Hospital /ID# 159450, Kochi
  - Hosoda Clinic /ID# 152978, Kofu
  - Hanada Internal Medicine Clin /ID# 155785, Koshigaya, Saitam
  - Cosmos Clinic /ID# 152298, Kōriyama
  - Ishida Medical Clinic /ID# 152297, Kōriyama
  - National Hosp Org Kumamoto /ID# 154783, Kumamoto
  - Seto Hospital /ID# 150056, Kumamoto
  - Kawasaki Medical School Hosp /ID# 152119, Kurashiki
  - Kurashiki Central Hospital /ID# 154656, Kurashiki
  - Mizushima Kyodo Hospital /ID# 152302, Kurashiki
  - Fukura Clinic /ID# 165273, Kurayoshi
  - National Hosp Org Kure Med Cen /ID# 152071, Kure, Hiroshima
  - Kurihara Central Hospital /ID# 152295, Kurihara
  - Kuroishi Hospital /ID# 153636, Kuroishi-aomori
  - Hori Internal Medicine Clinic /ID# 152291, Kushiro
  - Kyoto City Hospital /ID# 152188, Kyoto
  - Nakajima Clinic /ID# 157480, Kyoto
  - Aiseikai Yamashina Hospital /ID# 152100, Kyoto
  - Sawa Clinic /ID# 162881, Kyoto
  - NHO Kyoto Medical Center /ID# 152224, Kyoto
  - Otokoyama Hospital /ID# 153017, Kyoto
  - Kagawa University Hospital /ID# 154731, Kyoto
  - Machida Municipal Hospital /ID# 152184, Machida
  - Maebashi Red Cross Hospital /ID# 154707, Maebashi
  - Kagawa Rosai Hospital /ID# 152131, Marugame
  - Kono Naika clinic /ID# 152094, Marugame
  - Masuda Red Cross Hospital /ID# 153635, Masuda-shimane
  - Shinmatsudo Central General Ho /ID# 154668, Matsudo
  - Matsudo City Hospital /ID# 154666, Matsudo
  - Matsudo City Hospital /ID# 154764, Matsudo
  - Gibo Hepatorogy Clinic /ID# 154763, Matsumoto
  - Ehime Prefectural Central Hosp /ID# 154675, Matsuyama
  - Saiseikai Matsuyama Hospital /ID# 152270, Matsuyama
  - Tajiri Hospital /ID# 152320, Mimasaka
  - Kizawa Memorial Hospital /ID# 152096, Minokamo
  - Sumiyoshi Clinic Hospital /ID# 152093, Mito
  - Miyakonojo National Hospital /ID# 153007, Miyakonojō
  - Miyazaki Medical Center Hospit /ID# 152154, Miyazaki
  - Hepatopia Nishikohdai-naika /ID# 154788, Miyazaki
  - Haga Red Cross Hospital /ID# 152085, Mooka, Tochigi
  - Matsushita Memorial Hospital /ID# 154655, Moriguchi-shi
  - MC Ryokumeikai Yoshida Clinic /ID# 150055, Morioka
  - Abe Saien Clinic /ID# 153014, Morioka
  - Nagano Prefectural Kiso Hospit /ID# 152276, Nagano
  - Kimura Clinic /ID# 152146, Nagano
  - Tachikawa Medical Center /ID# 154784, Nagaoka
  - Jap Red Cross Nagasaki Genbaku /ID# 152300, Nagasaki
  - Jap Red Cross Nagasaki Genbaku /ID# 152303, Nagasaki
  - NHO Nagoya Medical Center /ID# 152294, Nagoya
  - Kita Hospital /ID# 158065, Nagoya
  - Japanese Red Cross Nagoya Daii /ID# 158099, Nagoya
  - Nakatsu Municipal Hospital /ID# 154673, Nakatsu
  - Kouseiren Namerikawa Hospital /ID# 154706, Namerikawa
  - Nara City Hospital /ID# 152189, Nara
  - Miyagiwa Internal Med Clinic /ID# 155887, Nara
  - Nara Prefectural Hospital /ID# 152234, Nara
  - Tani Internal Medicine Clinic /ID# 157448, Nayoro
  - Kameda Clinic /ID# 162879, Nishinomiya
  - Rinko Clinic /ID# 159449, Nishinomiya
  - Ooka Clinic /ID# 162880, Nishinomiya
  - Meiwa Hospital /ID# 152134, Nishinomiya, Hyogo
  - Noshiro Yamamoto Med. Assoc. /ID# 154785, Noshiro
  - Obihiro Dai-ichi Hospital /ID# 152238, Obihiro
  - Odawara Municipal Hospital /ID# 154761, Odawara
  - Eguchi Hospital /ID# 152292, Ogi
  - Okayama Saiseikai Outpatient Center Hospital /ID# 150057, Okayama
  - Kawaguchi Internal Medicine Cl /ID# 152301, Okayama
  - Heartlife Hospital /ID# 153619, Okinawa
  - Omuta City Hospital /ID# 152222, Omuta
  - Nishimura Clinic /ID# 154790, Omuta
  - Kita-harima Medical Center /ID# 153003, Ono
  - Onomichi Central General Hospi /ID# 152150, Onomichi
  - Tazuke Kofukai Foundation /ID# 152182, Osaka
  - Gokeikai Osaka Kaisei Hospital /ID# 153644, Osaka
  - Otemae Hospital /ID# 152987, Osaka
  - Center Clinic /ID# 161746, Osaka
  - Osaka Police Hospital /ID# 154781, Osaka
  - NTT WEST Osaka Hospital /ID# 157445, Osaka
  - Mori Clinic /ID# 157489, Osaka
  - Kansai Denryoku Hospital /ID# 155966, Osaka
  - Tamai Clinic /ID# 164951, Osaka
  - Osaka General Medical Center /ID# 160907, Osaka
  - Kansai Medical Univ Takii Hosp /ID# 152130, Osaka
  - Osaka Hospital /ID# 152168, Osaka
  - Asai Orthopedic /ID# 153015, Osaka
  - Osaka Gen Hosp West Railway /ID# 155962, Osaka
  - Tokai University Oiso Hospital /ID# 157456, Ōiso
  - Oita Red Cross Hospital /ID# 152289, Ōita
  - Oita Midical Center /ID# 154737, Ōita
  - Oita Prefectural Hospital /ID# 165261, Ōita
  - Mori Internal Medicine Clinic /ID# 157446, Ōita
  - Aso Shoukaki-naika /ID# 164142, Ōita
  - Ome Municipal General Hospital /ID# 153653, Ōme
  - Nasu Red Cross Hospital /ID# 152972, Ōtawara
  - Otsu City Hospital /ID# 152155, Ōtsu
  - Japanese Red Cross Otsu Shiga /ID# 153640, Ōtsu
  - Ryugasaki Saiseikai Hospital /ID# 153639, Ryūgasaki
  - Nakayama Medical Clinic /ID# 157481, Saga
  - Imari Arita Kyoritsu Hospital /ID# 152321, Saga
  - Saga Medical Center Koseikan /ID# 152989, Saga-shi, SAGA
  - Japanese Red Cross Sagamihara /ID# 153000, Sagamihara
  - Fuchinobe General Hospital /ID# 152996, Sagamihara
  - Sagamino Hospital /ID# 154676, Sagamihara
  - Saitama Citizens Medical Ctr /ID# 162882, Saitama
  - Honda Internal Clinic /ID# 157497, Saitama
  - Bellland General Hospital /ID# 152148, Sakai
  - Osaka Rosai Hospital /ID# 152286, Sakaishi
  - Nihonkai General Hospital /ID# 152973, Sakata-shi
  - Takayanagi Clinic /ID# 152975, Sakura
  - Hyogo-Chuo National Hospital /ID# 157441, Sanda
  - Hokkaido University Hospital /ID# 152982, Sapporo
  - IMS Sapporo Digestive Disease /ID# 154733, Sapporo
  - Sapporo Hokuyu Hospital /ID# 154709, Sapporo
  - Sasebo Chuo Hospital /ID# 154657, Sasebo
  - JR Sendai Hospital /ID# 152240, Sendai
  - Sendai Kousei Hospital /ID# 152181, Sendai
  - Sendai Red Cross Hospital /ID# 160908, Sendai
  - Shinmen Internal Medicine Clin /ID# 152172, Sennan
  - Tosei General Hospital /ID# 154710, Seto
  - NHO Shizuoka Medical Center /ID# 155897, Shimizu-sho
  - Shimonoseki Medical Center /ID# 165263, Shimonoseki
  - Dokkyo Medical University Hosp /ID# 152153, Shimotsuga
  - Dokkyo Medical University Hosp /ID# 153656, Shimotsuga
  - Anzunomori Clinic /ID# 157491, Shimotsuke
  - Saka General Hospital /ID# 153637, Shiogama-miyagi
  - Shobara Red Cross Hospital /ID# 156385, Shōbara
  - Saiseikai Suita Hospital /ID# 152171, Suita
  - Suita Municipal Hospital /ID# 153634, Suita-osaka
  - Konishi Medical Clinic /ID# 162886, Suzuka
  - Tachikawa Hospital /ID# 157458, Tachikawa
  - Gifu Prefectural Tajimi Hosp /ID# 152187, Tajimi
  - Takamatsu Red Cross Hospital /ID# 154711, Takamatsu
  - Kagawa Prefectural Central Hos /ID# 152293, Takamatsu
  - Sawada Hepatology & Gastro /ID# 157490, Takaraduka
  - Harano Internal Medicine Clini /ID# 154787, Takarazuka
  - Takarazuka City Hospital /ID# 152267, Takarazuka
  - Tenjin Tanaka Internal Medicin /ID# 162883, Takatsuki
  - Hamada Clinic /ID# 152142, Tatebayashi
  - Eastern Chiba Medical Center /ID# 155786, Togane, Chiba
  - Toki General Hospital /ID# 148821, Toki
  - Okubo Hospital /ID# 161751, Tokushima
  - Nihon University Hospital /ID# 159453, Tokyo
  - Mitsui Memorial Hospital /ID# 155891, Tokyo
  - The Jikei University Hospital /ID# 154671, Tokyo
  - Tokyo Takanawa Hospital /ID# 152133, Tokyo
  - kyo-wa Clinic /ID# 162884, Tokyo
  - The University of Tokyo Hospital /ID# 158069, Tokyo
  - Juntendo University Hospital /ID# 153555, Tokyo
  - Nippon Medical School Hospital /ID# 155787, Tokyo
  - Tobu Chiiki Hospital /ID# 155968, Tokyo
  - Tokyo Metropolitan Bokutoh Hos /ID# 152977, Tokyo
  - Tokyo Rinkai Hospital /ID# 152984, Tokyo
  - Shibata Hepatology Clinic /ID# 152141, Tokyo
  - Toshiba General Hospital /ID# 152161, Tokyo
  - Hojo Clinic /ID# 165271, Tokyo
  - Toho Univ Med Ctr Omori Hosp /ID# 153620, Tokyo
  - Ebara Hospital /ID# 154650, Tokyo
  - Mishuku Hospital /ID# 152136, Tokyo
  - Tokyo Yamate Medical Center /ID# 152284, Tokyo
  - Sato Gastro Med Clinic /ID# 154791, Tokyo
  - Tokyo Metropolitan Geriatric /ID# 153011, Tokyo
  - Juntendo Univ Nerima Hosp /ID# 152282, Tokyo
  - JP Red Cross Musashino Hosp /ID# 150052, Tokyo
  - NHO Tokyo Hospital /ID# 164132, Tokyo
  - Tonami General Hospital /ID# 152214, Tonami
  - Matsuda Internal Medicine Clin /ID# 152152, Tottori
  - Toyama Prefectural Ctr Hosp /ID# 152102, Toyama
  - Fujita Health University Hosp /ID# 156384, Toyoake
  - Toyohashi Municipal Hospital /ID# 153012, Toyohashi
  - Toyonaka Municipal Hospital /ID# 152299, Toyonaka
  - Ehime University Hospital /ID# 152273, Tōon
  - Mie Syokaki Clinic /ID# 158068, TSU, MIE
  - Sugiyama Clinic /ID# 161750, Tsukuba
  - University of Tsukuba Hospital /ID# 155784, Tsukuba
  - Tsuyama Chuo Hospital /ID# 154736, Tsuyama
  - Shizu Clinic /ID# 154766, Tsuyama
  - Yamaguchi University Hospital /ID# 153553, Ube
  - Shinshu Ueda Medical Center /ID# 153556, Ueda
  - Okinawa Prefectural Chubu Hosp /ID# 153006, Uruma
  - Sato Daiichi Hospital /ID# 154734, Usa
  - Saiseikai Utsunomiya Hospital /ID# 152974, Utsunomiya
  - Shinozaki Medical Clinic /ID# 159454, Utsunomiya
  - Seike Clinic /ID# 154765, Uwajima
  - Saiseikai Wakayama Hospital /ID# 153654, Wakayama
  - Wakayama Rosai Hospital /ID# 154732, Wakayama
  - Wakayama Medical University /ID# 155969, Wakayama
  - NHO Saitama National Hospital /ID# 153013, Wako
  - Gihoku Kosei Hospital /ID# 152158, Yamagata
  - Tohoku Central Hospital /ID# 152101, Yamagata
  - Gondo Medical Clinic /ID# 164952, Yame
  - Ishinkai Yao General Hospital /ID# 152983, Yao
  - Ushiroya Clinic /ID# 157443, Yashio
  - Kainan Hospital /ID# 154712, Yatomi-shi
  - Mie Prefectural General Medica /ID# 157442, Yokkaichi
  - Yokohama Rosai Hospital /ID# 154713, Yokohama
  - Hayashi Clinic /ID# 152143, Yokohama
  - Showa Univ Fujigaoka Hosp /ID# 153655, Yokohama
  - Oka Medical Clinic /ID# 154708, Yokohama
  - Shirato Clinic /ID# 154782, Yokohama
  - National Hosp Org Yokohama /ID# 159452, Yokohama
  - Yamauchi Internal Medicine Cli /ID# 154792, Yokosuka
  - Yamauchi Internal Medicine Cli /ID# 154793, Yokosuka
  - Josai Hospital /ID# 153009, Yūki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/ombitasvir_dasabuvir_P15-336.pdf